CLINICAL TRIAL: NCT03378050
Title: Efficacy and Feasibility of a Multi-component Individualized Telephone-based Support Intervention for Adult-child Caregivers Caring for Parents With Dementia in China: Study Protocol of a Randomized Controlled Trial
Brief Title: A Trial of a Multi-component Individualized Telephone-based Support Intervention for Adult-child Caregivers Caring for Parents With Dementia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Never Began
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Yu12.17
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: A randomized, controlled trial (RCT) will be used to compare a 12-week intervention group with a waiting-list control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a multi-component individualized support intervention "HEART", which will consist of 12 sessions in four stages.
  Interventions: Behavioral: HEART
- Control group (Active Comparator): Participants is the control group will be placed on a waiting list for 12 weeks. They will receive the intervention, after they complete the 12-week follow-up assessment. Caregivers in the control group will receive 12 week follow-up as usual (FU) including two brief "check-in" calls and an outcome measures call during the study period.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: HEART — The intervention group will receive a multi-component individualized support intervention "HEART", which will consist of 12 sessions in four stages. By using a comprehensive assessment targeting five components, an individualized intervention plan will be developed to address identified problems and unmet needs. Those five components consist of: Health, Emotion, Activities, Resources and Training.
  Arms: Intervention group
Other: Usual Care — Caregivers in the control group will receive 12 week follow-up as usual (FU) including two brief "check-in" calls and an outcome measures call during the study period.
  Arms: Control group

SUMMARY:
This is the first randomized controlled trial exploring the implementation of a multi-component individualized telephone-based support intervention for adult-child caregivers caring for parents with dementia in China. Results hold the potential to inform the further development of family caregiver supportive services.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the efficacy and feasibility of a multi-component individualized telephone-based support intervention (HEART) for adult-child caregivers caring for parents with dementia in China.

The primary hypothesis to test is whether the HEART is more efficacious in reducing caregiver burden than the follow-up as usual (FU) in dementia adult-child caregivers.

Secondary hypotheses include the following:

1. The HEART is more efficacious in improving health related quality of life than the FU in dementia adult-child caregivers.
2. The HEART is more efficacious in protecting reciprocal Filial Piety than the FU in dementia adult-child caregivers.
3. The HEART is more efficacious in relieving CR's behavioral and psychological symptoms of dementia (BPSD) than the FU in dementia adult-child caregivers.
4. The HEART group has a higher satisfaction with the intervention than the FU group.

In addition, two research questions will be answered by qualitative data from process evaluation for the feasibility of the HEART intervention. The research questions are as follows:

1. To what extent can the HEART intervention be delivered as planned?
2. What are the barriers to and facilitators of the HEART intervention?

ELIGIBILITY:
Inclusion Criteria:

* Primary caregivers being adult children (age 18 or older) who have spent at least 2 hours per day over the last 3 months caring for a parent with a diagnosis of dementia.
* Must have telephone access.
* Caregivers will not end their primary caregiving role within 6 months of study enrollment.

Exclusion Criteria:

* Cognitive impairment or intellectual disability.
* Those who are providing care for another relative with chronic physical or mental diseases.
* Pregnant women (Because it is unlikely that this group would be primary caregivers except in exceptional circumstances, the consideration of which was beyond the scope of this research).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Caregiver Burden | 12 weeks
  Caregiver burden will be assessed using the 12-item version of Zarit Burden Interview (12-item ZBI) to measure caregiver burden (Bédard, 2001; Zarit, 1980). Each item is rated on a 5-point Likert scale from 0 (never) though 4 (nearly always), yielding a possible range of 0 to 48. Higher scores indicate greater levels of caregiver burden. This short version and The Chinese version of 12-item ZBI has excellent internal consistency (Cronbachα= 0.87); and is highly correlated with the full measure (r = 0.952) (Lin, 2017; Wang, Yand, & Hou, 2006).

SECONDARY OUTCOMES:
Caregiver Burden | Baseline, 6 weeks and 24 weeks
  Caregiver burden will be assessed using the 12-item version of Zarit Burden Interview (12-item ZBI) to measure caregiver burden (Bédard, 2001; Zarit, 1980). Each item is rated on a 5-point Likert scale from 0 (never) though 4 (nearly always), yielding a possible range of 0 to 48. Higher scores indicate greater levels of caregiver burden. This short version and The Chinese version of 12-item ZBI has excellent internal consistency (Cronbachα= 0.87); and is highly correlated with the full measure (r = 0.952) (Lin, 2017; Wang, Yand, & Hou, 2006).
Health Related Quality of Life | Baseline, 6 weeks, 12 weeks and 24 weeks
  HRQoL will be measured using the 12-item Short Form Health Survey (SF-12), which is wildly used and has proved its feasibility in both self-administered and telephone interview (Lungenhausen et al., 2007; Ware Jr, Kosinski, & Keller, 1996). SF-12 consists of the mental component summary (MCS) and the physical component summary (PCS) with scores ranging from 0 to 100. Higher scores correspond to higher HRQoL. The Chinese version of SF-12 has been proved satisfactory for measuring and evaluating the quality of life for Chinese (Lam, Eileen, & Gandek, 2005).
Reciprocal Filial Piety | Baseline, 6 weeks, 12 weeks and 24 weeks
  The 8-item Reciprocal Filial Piety Scale (RFPS) (Yeh and Bedford, 2003) will used to measure RFP of adult children caring for their parents. This instrument uses a 5-point Likert scale from 1 (strongly disagree) to 6(strongly agree), yielding a total RFPS ranging from 8 to 48. Higher scores indicate greater RFP. Coefﬁcient (Cronbach) α for RFPS was 0.92, suggesting excellent reliability in this sample.
BPSD | Baseline, 6 weeks, 12 weeks and 24 weeks
  Caregivers' behavioral symptoms and caregivers' behavior-related reactions will be measured by the Neuropsychiatric Inventory Questionnaire (NPI-Q) (Kaufer et al., 2000), which covers 12 neuropsychiatric symptom domains. A "yes" or "no" screening question is used for each of the symptom. If the answer is "yes", caregivers are asked to rate the severity and distress of the symptoms in the last 4 weeks. The severity of the symptom is assessed in terms of on 3-point scale (1-mild, 2-moderate, 3-severe), yielding a possible range of 0 to 36. Caregiver distress associated with the symptom is rated by a 5-point Likert scale from 1 (mild) to 5(extreme), yielding a possible range of 0 to 60. The psychometric properties of English and Chinese versions are validated (Kaufer et al., 2000; Xie, Wang, & Yu, 2005).
Satisfaction with and benefits from the Intervention | 12 weeks and 24 weeks
  Caregivers will complete 8 questions about their satisfaction and benefits from participating in the study at the conclusion of the study. The measure uses a 5-point Likert scale from 1 (not at all) to 5(a great deal), yielding a total score ranging from 8 to 40.

IPD SHARING:
Plan to Share IPD: Undecided